CLINICAL TRIAL: NCT05339594
Title: Post-Market Clinical Follow-up Registry of Patients Requiring Nerve Gap Repair From Integra
Brief Title: REINVENT Registry (Registry of the Nerve Gap Repair From Integra)
Status: Terminated | Type: Observational
Why Stopped: Slow Enrollment, Sponsor Decision
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: T-INVENT-001
Record Dates: First submitted 2022-04-06; First posted 2022-04-21 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Nerve Injuries
Keywords: Digital Nerve Gap Repair
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- NeuraGen Nerve Guide: Integra NeuraGen nerve guide is an absorbable implant for the repair of peripheral nerve gaps.
  Interventions: Device: NeuraGen
- NeuraGen 3D Nerve Guide Matrix: Integra NeuraGen 3D Nerve Guide Matrix is a resorbable implant for the repair of peripheral nerve gaps.
  Interventions: Device: NeuraGen 3D

INTERVENTIONS:
Device: NeuraGen — NeuraGen nerve guide is an absorbable implant for the repair of peripheral nerve gaps.
  Groups: NeuraGen Nerve Guide
Device: NeuraGen 3D — NeuraGen 3D Nerve guide matrix is a resorbable implant for the repair of peripheral nerve gaps.
  Groups: NeuraGen 3D Nerve Guide Matrix

SUMMARY:
This is a prospective, multi-center, observational registry designed to evaluate two of Integra's collagen nerve gap repair products (NeuraGen® Nerve Guide and NeuraGen® 3D Nerve Guide Matrix). This registry will collect data on the outcome measures throughout the follow-up period for each patient. Data will be collected per standard of care.

DETAILED DESCRIPTION:
Integra NeuraGen Nerve Guide has been approved for clinical use since 2001 and has become a recognized clinical option for clinical nerve repair for the type of injuries evaluated in this registry. Integra NeuraGen Nerve Guide is used in this registry as a comparator to a next-generation advanced nerve guide, Integra NeuraGen 3D Nerve Guide Matrix, that is based on the original Integra NeuraGen Nerve Guide technology but contains a regenerative matrix in the lumen.

Centers chosen for participation will be current users of Integra's collagen nerve gap repair products listed above.

ELIGIBILITY:
Inclusion Criteria:

* Subject has undergone nerve gap repair utilizing NeuraGen or NeuraGen 3D
* Subject is willing and able to comply with postoperative procedures and visits such as immobilization, etc.
* Subject had a digital nerve injury that occurred up to 90 days prior to the nerve gap repair surgery detailed in this protocol.
* Subject had digital nerve injury(ies) that involve(s) complete nerve section of a sensory nerve of the palmar aspect of the hand that is distal to the palmer crease of the hand.
* Subject requires only a single repair per proper digital nerve branch

Exclusion Criteria:

* Subject has a known history of hypersensitivity to bovine-derived or chondroitin-based materials.
* Subject has participated in another clinical trial using an investigational drug or device within 30 days prior to the nerve repair surgery detailed in this protocol.
* Subject's hand injury is of a nature which could negatively impact healing of the target nerves such as a crush or avulsion injury, incomplete transection of the target nerve, or complete separation of the digit affiliated with the target nerve
* Subject has debris due to injury of the affected hand where contamination cannot be ruled out.
* Subject has pre-existing nerve lesions or known diagnosis of compressive neuropathy of median or ulnar nerves (i.e., Cubital or carpal tunnel syndrome)
* Subject has an infection of the area around the nerve defect.
* Subjects with diagnosed Peripheral Vascular Disease and Peripheral Arterial Disease
* Subject is known to have received immunosuppressive or antineoplastic agents or systemic steroids within 7 days of the study.
* Subject is known to have had or will require radiation or other therapy to the target hand or limb which may impact nerve healing.
* Subject has a history of injury to or a congenital abnormality of the target or contralateral hand or limb which may impact nerve healing or confound study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects with have had a repair of a peripheral nerve injury in the upper extremity distal to the palmer crease of the hand and without previous repairs.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
The primary clinical outcome measure is an evaluation of meaningful recovery as expressed by the Medical Research Council (MRC) scale as determined by the 2-point discrimination test (2PD). | 18 Months
  The primary endpoint success is when each subject reaches meaningful recovery, which is defined as an MRC score of S3+ or S4 (fair, good or excellent 2PD) of the pulp assessment of the distal phalanx of the affected digit(s).

SECONDARY OUTCOMES:
Evaluation of Static 2 Point Discrimination (s2PD) using DeMayo 2-point discrimination device | 18 Months
  To be assessed via in office visits
Evaluation of Moving 2PD using DeMayo 2-point discrimination device | 18 months
  To be assessed via in office visits
Evaluation of Michigan Hand and Outcomes Questionnaire (MHQ) | 15 Months
  To be assessed via web based tool during at home visits
Evaluation of Visual Analog Scale for Pain (VAS) | 15 Months
  To be assessed via web based tool during at home visits

CONTACTS AND LOCATIONS:
Overall Officials: Maria Leonard, BSN,RN,CTBS, Study Director — Integra LifeSciences
Locations (6):
- United States (6):
  - Indiana Hand to Shoulder Center, Indianapolis, Indiana
  - Washington University at St Louis, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia